CLINICAL TRIAL: NCT07114783
Title: Dual-function Semirigid Thoracoscopy Versus Rigid Thoracoscopy for the Diagnosis of Pleural Disease: a Randomised Controlled Trial
Brief Title: Dual-function Semirigid Thoracoscopy Versus Rigid Thoracoscopy for the Diagnosis of Pleural Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2025-UE-2
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-02

CONDITIONS: Pleural Effusion Disorder
Keywords: Medical Thoracoscopy; Pleural Disease
MeSH Terms: conditions — Pleural Effusion; Pleural Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-function Semi-rigid Thoracoscopy (Experimental)
  Interventions: Device: Dual-function semi-rigid thoracoscopy
- Rigid Thoracoscopy (Other)
  Interventions: Device: Rigid thoracoscopy

INTERVENTIONS:
Device: Dual-function semi-rigid thoracoscopy — Patients received pleural biopsy via dual-function semi-rigid thoracoscopy.
  Arms: Dual-function Semi-rigid Thoracoscopy
Device: Rigid thoracoscopy — Patients received pleural biopsy via rigid thoracoscopy.
  Arms: Rigid Thoracoscopy

SUMMARY:
Medical thoracoscopy (rigid and semirigid) is an effective, safe method for diagnosing and managing pleural diseases. Rigid thoracoscopy demonstrates superior overall diagnostic yield compared to semirigid techniques (flexible forceps/cryobiopsy) due to its ability to obtain larger, deeper biopsies with rigid forceps. However, diagnostic rates become similar when biopsies are successfully obtained.

Limitations of rigid thoracoscopy include restricted maneuverability (especially in posterior/mediastinal areas), increased procedural pain from leveraging against ribs and larger trocars, higher sedation requirements, and a steep learning curve for pulmonologists.

To address these issues, a novel dual-function semirigid thoracoscope (UE FET-680, China) was developed. Its straight working channel accommodates standard rigid biopsy forceps, potentially matching rigid thoracoscopy's diagnostic yield while improving usability. This randomized trial will compare the efficacy and safety of this new device versus conventional rigid thoracoscopy in undiagnosed exudative pleural effusions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Patients with unilateral pleural effusion of unclear aetiology after less invasive means of diagnosis;
3. Fully informed of the purpose and method of the study, agreed to participate in the study, and signed the informed consent form.

Exclusion Criteria:

1. Patients with PaO2/FiO2 <300;
2. Patients with a tendency for uncontrolled bleeding, unstable cardiovascular status or severe heart failure;
3. Patients with complete pleural symphysis, where it was not possible to create a pneumothorax, were excluded subsequently;
4. Patients with refractory cough;
5. Patients with Eastern Cooperative Oncology Group performance status 4;
6. Patients did not agree to participate in this study;
7. Participation in other studies within three months without withdrawal or termination will affect the observation of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 7 days after the procedure.
  Proportion of all individuals undergoing the diagnostic procedure under evaluation in whom a specific diagnosis is established based on the consensus definition.

SECONDARY OUTCOMES:
Complications incidence | 7 days after the procedure.
  The incidence of procedure-related complications.
Size of specimen | Day 7 after procedure
  Regarding biopsy size the total area is measured by the largest cross-sectional area under magnificence. Each sample was measured twice and the arithmetic mean of both measurements is accepted. All areas were calculated automatically and provided in mm2 by using ImageJ software (ImageJ, Marlyand, USA).
Quality of specimen | 7 days after procedure
  Biopsy quality was determined by tissue depth. A thoracoscopic biopsy specimen, including fatty tissue of the thoracic wall, was considered to be a deep biopsy and therefore of high quality.
Interpretability of the specimen | 7 days after procedure
  The interpretability of specimens is assessed as below:
  1. Easily interpretable: enough tissue with all elements required for diagnosis;
  2. Interpretability with some difficulty: less tissue or fewer diagnostic elements, diagnosis less reliable;
  3. Interpretable with great difficulty: little tissue or scant diagnostic elements, low reliability of diagnosis;
  4. Non-interpretable: diagnosis not possible.

OTHER OUTCOMES:
Procedural time | 1 day after procedure
  The procedural time was measured from incision to the final wound closure.
Pain degree | 1 day after procedure
  Pain was measured after the procedure with a VAS, ranging from no pain at all to worst possible pain.
Participant satisfaction | 1 day after procedure.
  Participant satisfaction was assessed with a Likert scale of 1 to 5, ranging from very dissatisfied to very satisfied.